CLINICAL TRIAL: NCT06983132
Title: Natural History of Familial Cerebral Cavernous Malformations: the CCM_Italia Cohort Study
Acronym: CCM_Italia
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other); Istituto Giannina Gaslini (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Azienda Ospedaliero-Universitaria Careggi (Other); University of Bari (Other); Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona (Other)
Responsible Party: Sponsor
Other Study IDs: ID 5417; PNRR-MR1- 2023-12378478 (Other Grant/Funding Number: Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan)
Record Dates: First submitted 2025-04-30; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-04

CONDITIONS: CCM; Familial Cerebral Cavernous Malformation
Keywords: CCM; fCCM
MeSH Terms: conditions — Familial cerebral cavernous malformation | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — 15,5 ml of blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with symptomatic and asymptomatic familial cerebral angiomatosis will be included.: Patients with symptomatic and asymptomatic familial cerebral angiomatosis will be included. Subjects without genetic diagnosis will not be included. Other exclusion ctiteria will be current inclusion in a different clinical study, inability to cooperate with study procedures, contraindication to cerebral MRI.
  Interventions: Diagnostic Test: Cerebral imaging (MRI) according to a dedicated protocol with central MRI reading; Diagnostic Test: Determination of circulating biomarkers

INTERVENTIONS:
Diagnostic Test: Cerebral imaging (MRI) according to a dedicated protocol with central MRI reading — Cerebral MRI according to dedicated protocol, central MRI reading.
  Other Names: Circulating biomarkers; Cerebral MRI
Diagnostic Test: Determination of circulating biomarkers — High-throughput molecular analysis will be performed on plasma samples collected assessing a selected panel of biomarkers, associated with endothelial cell profiles using automated and high-throughput ELISA. The interactions between mutation profile, protein biomarkers, and clinical variables will be correlated with patients' outcomes.

SUMMARY:
Patients with symptomatic and asymptomatic familial cerebral cavernous malformation (fCCM) will be included. The goal of this observational study is to learn about the long-term evolution of this condition. The subjects enrolled will be followed for two years and will undergo an annual neurological examination with the recording of clinical events, a brain MRI according to a dedicated protocol, and a blood draw for the determination of circulating biomarkers. They will also be asked to complete questionnaires on quality of life. The data derived from the study will allow for a better understanding of the natural history of the disease and the identification of neuroradiological and/or circulating biomarkers capable of predicting the clinical evolution of the condition.

DETAILED DESCRIPTION:
CCM_Italia is an observational non interventional national multicentric registry.

Patients will be enrolled prospectively and followed for a 2 years period through annual neurological evaluation, cerebrale MRI according to dedicated protocol (central reading) and blood sample to assess circulating biomarkers.

The study has been funded by National Recovery and Resilience Plan.

In the contest of the present study, pediatric and adult patients affected by genetically confirmed fCCM will be enrolled according to the inclusion and exclusion criteria which have been developed to include a large number of fCCM patients, representative of the heterogeneity of fCCM disease, spanning from the asymptomatic to the high-risk cases.

This registry is primarily designed to collect real-world data without influencing or interfering with the standard clinical practice and external monitoring is not planned. Since the data collection process is passive and observational by nature, the risk to patient safety and data integrity is minimal compared to interventional studies. Internal data quality controls and oversight mechanisms are planned. The use of standardized protocols for data entry ensures consistency across all entries. This reduces variability caused by different personnel and minimizes errors in recording patient information, pathology findings, and other relevant data. We plan periodic audits of the registry data helps identify discrepancies, incomplete records, or inconsistencies. Cross-checking data entries against source documents or original reports will minimize data loss.

A comprehensive training for staff responsible for data entry ensures they understand the data standards and procedures. Certifying personnel helps maintain high levels of accuracy and consistency over time. Inter-observer reliability among neuroradiologist in charge of imaging analysis ensures consistency in data collection. A constant feedback from users and data contributors encourages reporting of issues or inconsistencies, fostering ongoing improvements to data quality processes.

• Study procedures The quality assurance of the study is maintained through regular training sessions and periodic online meetings. These initiatives ensure consistent protocols are followed across all team members, promoting uniformity in patient enrollment and data collection. Specifically, training sessions provide comprehensive guidance on study procedures and data entry standards, while scheduled online meetings allow for ongoing monitoring, clarification of any issues, and reinforcement of best practices. This continuous educational approach helps to minimize variability, ensuring that patient recruitment and data collection within the REDCap database are accurate, reliable, and standardized throughout the study duration.

In accordance with clinical practice, annual cerebral MRI will be performed in the Neuroradiology Unit of the referral hospital preferably on the same day as the clinical assessment, otherwise planned within 1 month for inclusion visit/+/- 40 days for follow-up visit (T0-T1-T2). The MRI protocol will include: sagittal 3D T1¬weighted turbo field echo, sagittal 3D T2¬weighted turbo spin echo, sagittal 3D fluid¬ attenuated inversion recovery, axial diffusion¬ weighted imaging, axial sus-ceptibility ¬weighted imaging, and axial T2¬weighted gradient echo. The current protocol is in line with normal clinical practice. The collected MRIs will be assessed centrally in the MRI core lab at Fondazione Cà Granda by blinded personnel. The following variables will be collected: different vascular lesion characteristics such as number, pattern and size of CCMs, signs of bleeding (Za-bramski classification) and number of the novo lesions. Advanced MRI techniques such as Quantitative Susceptibility Mapping, which is not routinely performed in the follow-up of CCM patients, will be applied and performed centrally at Fondazione Cà Granda in the MRI core lab to assess iron deposition and vessel permeability if available in the centre.

The uniformity of the MRI protocol is ensured through dedicated training sessions and the sharing of representative examinations. These measures serve to verify the correctness of the settings and ensure the comparability of the scans across different centers. Additionally, centralized image reading further strengthens the robustness of the project by maintaining consistent interpretation standards and reducing inter-observer variability. This comprehensive approach enhances the overall quality and reliability of the imaging data.

Besides the "standard" annual clinical assessment as described above, adult patients will annually be asked to complete specific questionnaires for Patient Reported Outcome Measures (PROMs) and Patient Reported Experience Measures (PREMs). These include the following standardized ques-tionnaires for depression: Beck Depression Inventory-II (BDI-2); Anxiety: Stait-Trait Anxiety Inventory X1 & X2 (STAI X-1 & STAI X-2) and Quality of Life: the Short Form 36 (SF-36), split into the physical and mental component scales (PCS and MCS).

Moreover in addition to the "standard" annual clinical assessment, patients will undergo blood sample collec-tion at the same moment as their annual clinical visit. Three vials, a total of 15.5 ml of blood will be collected in the outpatient clinic of the referral hospital.

All patients' clinical and radiological data as well as outcomes of questionnaires and specific information on clinical events will be de-identified and recorded on electronic case report files on the RedCap platform.

Blood samples (15,5 ml) will be collected during the clinical visits at baseline (T0) 12 months (T1) and 24 months (T2), according to specific standard operating procedures that will be shared by the biobank with all clinical centers participating in the study. Blood and plasma aliquots will be temporarily stored at -70°C at the local clinical centers until shipment in dry ice to the SATURNE biobank at IRFMN in Milan. The samples will be de-identified with a unique 6-digit code and centralized to the "Saturne" Biobank at IRFMN (certified UN EN ISO 9001:2015) for long-term storage in -70°C freezer under controlled condition for further analysis.A part of plasma samples will be used for analysis of biomarkers related to inflammation, coagula-tion, angiogenesis (such as C-reactive protein, PTX3, LBP, ROBO4, Tissue Factor, Endoglin, Thrombomodulin, CCL5, CXCL-4) performed at Policlinico di Bari. These biomarkers will be measured by enzyme-linked immunosorbent assay (ELISA) or using enzymatic-colorimetric and immunoturbidimetric method (i.e. CRP). Remaining aliquots not used for the analyses present in the protocol will be stored in the biobank and will be used for future studies to identify new biomarkers of interest of CCM.

• Sample size and statistical analysis The primary objective is to evaluate the new occurrence of CCM-related clinical events in patients with fCCM. CCM-related clinical events, the primary endpoint, are defined as intra-cerebral hemor-rhage (ICH) and focal neurological deficits (FND).

The primary endpoint, new occurrence of CCM-related clinical events, defined as intra-cerebral hemorrhage (ICH) and focal neurological deficits (FND), excluding seizures, are expected in about 5.6% of the population based on the Treat_CCM trial (1). Assuming that 5,6% of the subjects in the population will develop an CCM-related clinical event within the CCM_Italia cohort, we need to include at least 100 patients (including a dropout of 8%) for estimating this expected proportion with 95% confidence and 4,7% absolute precision.

Furthermore, it can be shown that including 100 patients with fCCM allows to obtain sufficient power (equal to 80%) to evaluate the secondary endpoint. Once a patient cohort has been created which includes a long-term standardized follow-up of patients, we can leverage this cohort to assess potential biomarkers to monitor disease activity, aim 2. Hypothetically, a cohort with at least 100 patients will allow us to have enough power to detect a minimal hazard ratio of 2.15 for identifying patients with increased disease activity (defined as CCM-related adverse events or the development of at least 5 new CCM lesions during the two years of observation). The Treat_CCM study indicat-ed that 55% of the fCCM patients will experience increased disease activity. Dividing the popula-tion by the median level of a biomarker of interest (thus obtaining 2 groups of 50 persons) would give us a statistically significant result if the HR of this biomarker is at least 2.15 (power 80% and alpha 0.05) (4,5). This was assessed by means of R, using function ssizeEpi.default (Library Pow-erSurvEpi): power 80%, p=0.5 (population split 50/50 by median biomarker level), psi=0.55 (55% experienced increased disease activity in Treat_CCM), rho2= 0.025025 (based upon the correlation of CXCL4 with disease activity in the Treat_CCM cohort), alpha 0.05, theta 2.15.Baseline characteristics will be presented for the total population and by relevant characteristics (i.e. sex, age classes, number of CCM lesions). Baseline subgroups will be compared by descriptive uni-variate statistics.

1. Primary endpoint: Patient characteristics will be compared by means of descriptive analyses to assess patients with clinical events.
2. Secondary Endpoints:

   1. Clinical secondary endpoints: individual components of the primary endpoint, ICH or FND, and other clinical secondary end-points such as seizures, headache or hospitalization will be assessed by means of descriptive anal-yses. In addition, Kaplan Meier curves will be constructed to illustrate the occurrence of clinical events over time.
   2. Biomarkers: in order to reach aim 2, assess biomarkers for the management of fCCM, Cox proportional hazards regression analyses will be performed to assess which circulating biomarkers are independently as-sociated with increased disease activity (defined as CCM-related adverse events or the development of at least 5 new CCM lesions during the two years of observation). All outcomes will be reported including a 95% confidence interval.
   3. Questionnaires: Global cognitive functioning, depression, anxiety and health related quality of life will be assessed at multiple time points and any changes over time will be described and assessed by repeated measures ANOVA.
   4. Imaging: Different vascular lesion characteristics, measured by MR imaging will be assessed for the total population and by relevant characteristics (i.e. sex, age classes, number of CCM lesions, etc). The evolution of MRI markers such as number of new lesions and size of lesions will be described and changes over time will be assessed by repeated measures ANOVA. The assessment of changes over time will be performed for all patients included in the cohort as change from baseline to 2 year follow-up.

Implementation of Standard Operating Procedures (SOPs) for our registry is essential for ensuring consistency, quality, and compliance in registry operations and analysis activities. Firstly, SOPs for patient recruitment help standardize eligibility criteria, recruitment strategies, and consent processes, thereby maximizing efficiency and ensuring ethical standards are maintained. Clear shared guidelines on data collection and data management are likely to ensure data accuracy, completeness, and confidentiality throughout the registry lifecycle.

Using Standard Operating Procedures (SOPs) for imaging data collection ensures consistency across different centers. SOPs provide detailed, standardized protocols that all sites follow, minimizing variability in how images are acquired. This uniformity is crucial for reliable comparison and analysis of imaging data, as it reduces discrepancies caused by differences in equipment settings, patient positioning, or imaging techniques. By adhering to SOPs, centers can maintain high-quality, reproducible data, which enhances the validity of multi-center studies and facilitates accurate interpretation of results.

The impact of missing data will be minimized through data collection protocols to reduce missingness, such as follow-up queries or alternative data sources.

ELIGIBILITY:
Inclusion Criteria:

* Patients with familial cerebral cavernous malformations (FCCM), documented by mutations in the CCM1, CCM2, or CCM3 genes;
* Asymptomatic patients or those with a history of clinical symptoms or events, such as intracerebral hemorrhage, stroke, permanent or transient focal deficits, seizures, disability, or any other neurological symptom presumably related to CCM;
* Life expectancy at least equal to the duration of the study follow-up;
* Written informed consent from the patient (or guardian in the case of minors) to participate in the study.

Exclusion Criteria:

* Implanted pacemaker or any other condition that precludes magnetic resonance imaging;
* Participation in another ongoing interventional clinical study;
* Inability to cooperate with the study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with familial cerebral cavernous malformations (FCCM), documented by mutations in the CCM1, CCM2, or CCM3 genes. Either symptomatic or asymptomatic subjects will be considered for inclusion
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Occurrence of CCM-related clinical events | 24 months
  New occurrence of intracerebral haemorrhage (ICH) or focal neurological deficits (FNDs)

SECONDARY OUTCOMES:
Other clinical manifestations | 24 months
  To evaluate the occurrence of seizure episodes and other CCM-related clinical events such as recurrent headaches.
Neuroradiological markers of disease progression | 24 months
  To identify neuroradiological markers of disease progression
  * CCM lesions (number)
  * CCM new lesions (number)
  * Location of lesions (number of CCM lesions in each of the following site: cerebellum, brainstem, basal ganglia and thalami, right cerebral hemisphere, left cerebral hemisphere)
  * Radiological characteristics (number of CCM lesions classified according to Zabramski classification: type I, II, III and IV ( Zabramski JM et al. J. Neurosurg. 1994 doi:10.3171/jns.1994.80.3.0422)).
Circulating biomarkers | 24 months
  To identify circulating biomarkers to predict clinical evolution and haemorrhagic risk sCD14 (ng/mL), LBP (ng/mL), ICAM-1 (ng/mL), VCAM-1 (ng/mL), ANG2 (pg/mL), sENG (pg/mL), CCL5 (ng/mL), THBS1 (ng/mL), CXCL4 (ng/ml), sROBO4 (pg/mL), TM (pg/mL), Tissue factor (pg/mL), cholesterol (mg/dL), HDL (mg/dL), Triglycerides (mg/dL), CRP (mg/L), PTX3 (ng/mL)

OTHER OUTCOMES:
Patients reported outcome measures | 24 months
  To assess overall cognitive function, disability, and perceived quality of life in patients with fCCM.
  Depression assessed by means of the Beck Depression Inventory-II (BDI-II). This scale allows us to distinguish the following levels of depression: score 0-9 no depression; score 10-18 slight depression; score 19-29 moderate depression; score 30-63 severe depression. Patients will be classified as depressed with a cutoff of 10.
  * Anxiety assessed by means of the Short Form Health Survey (forms X-1 and X-2, STAI X-1 and STAI X-2). A patient is classified as being in a state of anxiety while completing thequestionnaire if (s)he scores in the top 99% (for male individuals, this corresponds to a score of ≥65 and for female ≥62).
  * QoL assessed by means of the SF-36. A higher score indicates a better QoL.

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Policlinico di Bari, Bari
  - Careggi Hospital, Firenze, Florence
  - Istituto Giannina Gaslini, Genova, Genova
  - Fondazione IRCCS Cà Granda, Ospedale Maggiore Policlinico, Milan, Italy, Milan
  - Istituto di Ricerche Farmacologiche Mario Negri, Milan
  - San Giovanni di Dio e Ruggi d'Aragona", Salerno, Salerno

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Latouche A, Porcher R, Chevret S. Sample size formula for proportional hazards modelling of competing risks. Stat Med. 2004 Nov 15;23(21):3263-74. doi: 10.1002/sim.1915. PMID 15490425
- [Background] Schoenfeld DA. Sample-size formula for the proportional-hazards regression model. Biometrics. 1983 Jun;39(2):499-503. PMID 6354290
- [Background] Meessen JMTA, Abete-Fornara G, Zarino B, Castori M, Tassi L, Carriero MR, D'Alessandris QG, Al-Shahi Salman R, Blanda A, Nicolis EB, Novelli D, Caruana M, Vasami A, Lanfranconi S, Latini R. Patient-reported outcome measures in patients with familial cerebral cavernous malformations: results from the Treat_CCM trial. Front Neurol. 2024 Feb 14;15:1338941. doi: 10.3389/fneur.2024.1338941. eCollection 2024. PMID 38419711
- [Background] Lazzaroni F, Meessen JMTA, Sun Y, Lanfranconi S, Scola E, D'Alessandris QG, Tassi L, Carriero MR, Castori M, Marino S, Blanda A, Nicolis EB, Novelli D, Calabrese R, Agnelli NM, Bottazzi B, Leone R, Mazzola S, Besana S, Catozzi C, Nezi L, Lampugnani MG, Malinverno M, Grdseloff N, Rodel CJ, Rezai Jahromi B, Bolli N, Passamonti F, Magnusson PU, Abdelilah-Seyfried S, Dejana E, Latini R. Circulating biomarkers in familial cerebral cavernous malformation. EBioMedicine. 2024 Jan;99:104914. doi: 10.1016/j.ebiom.2023.104914. Epub 2023 Dec 18. PMID 38113759
- [Background] Lanfranconi S, Scola E, Meessen JMTA, Pallini R, Bertani GA, Al-Shahi Salman R, Dejana E, Latini R; Treat_CCM Investigators. Safety and efficacy of propranolol for treatment of familial cerebral cavernous malformations (Treat_CCM): a randomised, open-label, blinded-endpoint, phase 2 pilot trial. Lancet Neurol. 2023 Jan;22(1):35-44. doi: 10.1016/S1474-4422(22)00409-4. Epub 2022 Nov 17. PMID 36403580
- [Derived] Lanfranconi S, Scola E, Novelli D, Poggesi A, Pescini F, Pavanello M, Romano F, D'Alessandris QG, Marani W, Signorelli F, Iaconetta G, Torelli G, Fainardi E, Severino M, Remore LG, Bertani GA, Conte G, Capra V, Vasami A, Nicolis E, Contino G, Ronchi D, Palmieri MC, Previtali A, Mattogno PP, Sturiale CL, Solarino ME, Caliulo R, Bozzi MT, Fratini F, Zanier ER, Latini R, Meessen JMTA, Locatelli M; and the CCM_Italia investigators. Natural history of familial cerebral cavernous malformations: the CCM_Italia cohort study. Front Neurol. 2026 Jan 5;16:1668098. doi: 10.3389/fneur.2025.1668098. eCollection 2025. PMID 41561324